CLINICAL TRIAL: NCT05951998
Title: Frequency and Risk Factors of H.Pylori Infection in Children Presented by Dyspeptic Symptoms in Assiut University Children Hospital
Brief Title: Frequency of h.Pylori in Children With Dyspeptic Symptoms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Samy Fayek, principal investigator, Assiut University
Other Study IDs: H.pylori infection in children
Record Dates: First submitted 2023-04-10; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: H.Pylori Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The current work aim to:

Estimation of prevalence, Estimation of risk factors, Estimation of endoscopic picture of H. pylori infection in children presented with chronic or recurrent dyspeptic symptoms and/or non variceal hematemesis.

DETAILED DESCRIPTION:
Helicobacter pylori infection is a common problem in pediatric practice, it's an important cause of gastrointestinal pathology in children and its acquisition is related with poor socioeconomic conditions. H.pylori is a spiral, microaerophilic, gram-negative bacterium with four to six unipolar sheathed flagella.The human stomach, especially the antrum, is the most common reservoir of this agent. American board of orthodontists antibody blood group and Lewis blood-group antigen might expose cases to H. pylori infection, the most likely mode of transmission is fecal-oral or oral-oral. H.pylori infection is predominantly acquired during early childhood .

The majority of children with are asymptomatic although a percentage of the infected children develop H. pylori associated diseases such as iron deficiency anemia, B12 deficiency, chronic thrombocytopenic purpura. It can manifest with burning pain in the stomach, nausea, loss of appetite, bloating, weight loss.

Previous studies showed that geographic area, age, race, educational level, sanitation, and socioeconomic status are among the factors that influence the prevalence of H. pylori infection . No gender differences were found in the prevalence of H. pylori infection, while it was much higher among white people.

The overall prevalence of H. pylori infection in Egyptian school children was 72.38%. There was no significant difference in the prevalence of infection between boys and girls (73.80% vs. 70.34% respectively, or in the independent effect of sex by age. Of school children living in Sohag, 96.7% tested positive for H. pylori, compared with 81.3% of children from Giza and 61.9% from Cairo. Prevalence was also highest among children of low socio-economic class and decreased gradually among children of medium to high socio-economic class.

In a previous study conducted by Hunt et al., the prevalence of H. pylori was reported to be 48% among 2-4-year-old children in Ethiopia, while in Nigeria and Mexico it was 82% and 43%, respectively, among 5-9-year-old children..

The endoscopic findings in order of decreasing frequency in the Pediatric group were nodularity (93.0%), mucosal swelling (32.6%), spotty redness (25.6%), diffuse redness (18.6%), atrophy (9.3%), enlarged fold (4.7%), depressive erosion (4.7%), foveolar-hyperplastic polyp (2.3%), patchy redness (2.3%), red streak (2.3%), and raised erosion (2.3%).

Invasive and non-invasive tests could be used for diagnosis, while the gold standard is a biopsy specimen of gastrointestinal tract.

Triple therapy is considered to be the standard treatment for children. Proton pump inhibitor combined with two antibiotics has been shown to be very effective in clearing H. pylori from the stomach, it is recommended to treat with amoxicillin, clarithromycin and a proton pump inhibitor for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children from age of 3 years to age of 18 years.
* Children presented with chronic or recurrent dyspeptic symptoms(epigastric pain, post prandial fullness, early satiety, bleaching, heart burn ,bloating ,flatulence ,regurgitation ,nausea ,vomiting and/or halitosis) and/or non variceal hematemesis.

Exclusion Criteria:

* Children less than 3 years and more than 18 years.
* Children with variceal hematemesis.

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 100 child aged 3years to 18 years with H.pylori infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of frequency of H.pylori infection | Baseline
  2.Estimation of prevalence of H.pylori infection
  3.Estimation of risk factors of H.pylori infection
  4.Estimation of endoscopic picture of H. pylori infection in children presented with chronic or recurrent dyspeptic symptoms and/or non variceal hematemesis.

CONTACTS AND LOCATIONS:
Overall Officials: Gamal A Askar, Prof, Principal Investigator — Assiut University; Ashraf M Elsaghier, Prof, Principal Investigator — Assiut University